CLINICAL TRIAL: NCT06002750
Title: The Third People's Hospital of Hangzhou
Brief Title: Evaluation of Tp-e Interval and Tp-e/QT Ratio in Dermatomyositis and Analysis of Their Relationship With Inflammation
Status: Completed | Type: Observational
Sponsor: The Third People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Ling Pin, Chief physician, The Third People's Hospital of Hangzhou
Other Study IDs: 2021KA048
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Dermatomyositis; Myocardial Repolarization; Inflammation
MeSH Terms: conditions — Dermatomyositis; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dermatomyositis patients
  Interventions: Other: disease
- The control group was comprised of age- and gender-matched healthy volunteers

INTERVENTIONS:
Other: disease — Do you have dermatomyositis
  Groups: Dermatomyositis patients

SUMMARY:
The goal of this observational study is to investigate ventricular repolarization utilizing Tp-e intervals and Tp-e/QT ratios in patients with DM. The main questions it aims to answer are:

* 1.Exploring the changes in ventricular repolarization parameters (QT interval, QTc interval, QTd, Tp-e interval, Tp-e/QT ratio) in patients with dermatomyositis, providing quantifiable indicators for early detection of arrhythmia in dermatomyositis patients;
* 2.Exploring the role of inflammation in ventricular repolarization in DM patients, providing a basis for in-depth research on the diagnosis and prevention of arrhythmia in DM patients.

ELIGIBILITY:
Inclusion Criteria:

Regardless of gender, registered residence and education level, voluntarily participate in this study and sign the informed consent form.

Clinical diagnosis of Dermatomyositis.

Exclusion Criteria:

Previous history of heart disease (such as myocardial infarction, cardiac pacing, congenital heart disease, ischemic heart disease, etc.), chronic kidney disease, etc; Patients with other connective tissue diseases; Pregnant and lactating women.

Taking drugs that affect electrocardiogram indicators, such as macrolides, quinolones, quinidine, amiodarone, antipsychotic drugs, etc.

Patients with severe lack of case data.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dermatomyositis patients from November 2011 to November 2022 who visited our hospital, and a healthy control group consisting of the same number of gender and age matched healthy adults in a physical examination center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
QTc, Tp-e interval, and Tp-e/QT ratio were increased in DM patients. | November 2011 to November 2022
the Tp-e interval and Tp-e/QT ratio were positively correlated with Inflammation. | November 2011 to November 2022

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Hangzhou, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundberg IE. Expert Perspective: Management of Refractory Inflammatory Myopathy. Arthritis Rheumatol. 2021 Aug;73(8):1394-1407. doi: 10.1002/art.41762. Epub 2021 Jun 29. PMID 33844450
- [Background] Zhao L, Wang Q, Zhou B, Zhang L, Zhu H. The Role of Immune Cells in the Pathogenesis of Idiopathic Inflammatory Myopathies. Aging Dis. 2021 Feb 1;12(1):247-260. doi: 10.14336/AD.2020.0410. eCollection 2021 Feb. PMID 33532139
- [Background] Schwartz T, Diederichsen LP, Lundberg IE, Sjaastad I, Sanner H. Cardiac involvement in adult and juvenile idiopathic inflammatory myopathies. RMD Open. 2016 Sep 27;2(2):e000291. doi: 10.1136/rmdopen-2016-000291. eCollection 2016. PMID 27752355
- [Background] Kors JA, Ritsema van Eck HJ, van Herpen G. The meaning of the Tp-Te interval and its diagnostic value. J Electrocardiol. 2008 Nov-Dec;41(6):575-80. doi: 10.1016/j.jelectrocard.2008.07.030. PMID 18954608
- [Background] Antzelevitch C, Sicouri S, Di Diego JM, Burashnikov A, Viskin S, Shimizu W, Yan GX, Kowey P, Zhang L. Does Tpeak-Tend provide an index of transmural dispersion of repolarization? Heart Rhythm. 2007 Aug;4(8):1114-6; author reply 1116-9. doi: 10.1016/j.hrthm.2007.05.028. Epub 2007 Jun 8. No abstract available. PMID 17675094
- [Background] Naaraayan A, Meredith A, Nimkar A, Arora G, Bharati R, Acharya P. Arrhythmia prevalence among patients with polymyositis-dermatomyositis in the United States: An observational study. Heart Rhythm. 2021 Sep;18(9):1516-1523. doi: 10.1016/j.hrthm.2021.05.029. Epub 2021 May 26. PMID 34048962
- [Background] Indraratna P, Tardo D, Delves M, Szirt R, Ng B. Measurement and Management of QT Interval Prolongation for General Physicians. J Gen Intern Med. 2020 Mar;35(3):865-873. doi: 10.1007/s11606-019-05477-7. Epub 2019 Oct 25. PMID 31654357
- [Background] Korsholm SS, Andersson DC, Knudsen JB, Dastmalchi M, Diederichsen ACP, Gerke O, Witting N, Jacobsen S, Pecini R, Friis T, Krogager ME, Lundberg IE, Diederichsen LP. Myositis-specific autoantibodies and QTc changes by ECG in idiopathic inflammatory myopathies. Rheumatology (Oxford). 2022 Oct 6;61(10):4076-4086. doi: 10.1093/rheumatology/keac013. PMID 35048961
- [Background] Mendez Hernandez R, Ramasco Rueda F. Biomarkers as Prognostic Predictors and Therapeutic Guide in Critically Ill Patients: Clinical Evidence. J Pers Med. 2023 Feb 15;13(2):333. doi: 10.3390/jpm13020333. PMID 36836567
- [Background] Lazzerini PE, Capecchi PL, El-Sherif N, Laghi-Pasini F, Boutjdir M. Emerging Arrhythmic Risk of Autoimmune and Inflammatory Cardiac Channelopathies. J Am Heart Assoc. 2018 Nov 20;7(22):e010595. doi: 10.1161/JAHA.118.010595. No abstract available. PMID 30571503